CLINICAL TRIAL: NCT05972135
Title: Outpatient Administration of Teclistamab or Talquetamab for Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM165
Record Dates: First submitted 2023-07-12; First posted 2023-08-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Teclistamab (TECVAYLI™); Humanized IgG-4 PAA bispecific antibody; CD3 receptor complex; RRMM-Relapsed or Refractory Multiple Myeloma; MM-Multiple Myeloma; Tocilizumab prophylaxis; CRS- Cytokine Release Syndrome; Neurologic toxicity; ICANS-Immune Effector Cell-associated Neurotoxicity Syndrome; Talquetamab (TALVEY™); GPRC5D; BCMA; Oral dexamethasone prophylaxis
MeSH Terms: conditions — Multiple Myeloma; Cytokine Release Syndrome | interventions — talquetamab; tocilizumab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Teclistamab/Tocilizumab (Experimental): Participants will receive step up dosing of Teclistamab following the recommended dosage of TECVAYLI™ USPI followed by weekly dosing for twelve 28-day cycles, until disease progression, unacceptable toxicity, or the EOT (end of Cycle 12). Teclistamab dosing may be reduced to once every 2 weeks for participants who achieve partial response (PR) or better after 6 months of therapy.
  Interventions: Drug: Teclistamab; Drug: Tocilizumab
- Talquetamab/Tocilizumab (Experimental): Participants will receive step up dosing of Talquetamab following the recommended dosage of TALVEY™ USPI followed by every 2 week dosing for six 28-day cycles, until disease progression, unacceptable toxicity, or the EOT (end of Cycle 6). Talquetamab dosing may be reduced to once every 4 weeks for participants who achieve very good partial response (VGPR) or better after Cycle 4. Participants in the talquetemab arm cannot be re-screened for or re-enrolled into the teclistamab arm.
  Interventions: Drug: Talquetamab; Drug: Tocilizumab
- Teclistamab/Oral Dexamethasone (Experimental): Participants will receive step-up dosing of Teclistamab followed by weekly dosing for two cycles, every other week during Cycles 3-6 and once every 4 weeks from Cycles 7 through 12 until disease progression, unacceptable toxicity, or the EOT (end of Cycle 12). Teclistamab dosing may be reduced to once every 4 weeks for participants who achieve very good partial response (VGPR) or better starting with Cycle 3.
  Interventions: Drug: Teclistamab; Drug: Oral Dexamethasone

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered subcutaneously at step-up doses on Day 1, Day 4 and Day 8, one week after first treatment dose and weekly thereafter. In participants who have a partial response (PR) or better after 6 months of therapy, dosing frequency may be reduced to every 2 weeks.
  Other Names: (TECVAYLI™)
  Arms: Teclistamab/Oral Dexamethasone; Teclistamab/Tocilizumab
Drug: Talquetamab — Talquetamab will be administered subcutaneously at step-up doses on Day 1, Day 4, Day 8 and Day 15, one week after first treatment dose and every 2 weeks thereafter. In participants who have a very good partial response (VGPR) or better after Cycle 4, dosing frequency may be reduced to every 4 weeks
  Other Names: TALVEY™
  Arms: Talquetamab/Tocilizumab
Drug: Tocilizumab — Tocilizumab will be administered as a pretreatment medication in advance of administration of the first step-up dose of teclistamab or talquetamab on Cycle 1 Day 1.
  Other Names: Actemra
  Arms: Talquetamab/Tocilizumab; Teclistamab/Tocilizumab
Drug: Oral Dexamethasone — Oral dexamethasone will be administered as a pretreatment medication every 12 hours in 3 doses (PM/AM/PM) following each step-up dose and the first full dose of teclistamab in Cycle 1. A total of 9 doses of oral dexamethasone will be administered.
  Other Names: Decadron
  Arms: Teclistamab/Oral Dexamethasone

SUMMARY:
This is a phase II study to evaluate the outpatient administration of Teclistamab or Talquetamab in Multiple Myeloma patients

DETAILED DESCRIPTION:
* This is a three-arm, non-randomized, multicenter, prospective study in adult patients with RRMM, who are administered Teclistamab (TECVAYLI™) or Talquetamab (TALVEY™), in the post-marketing setting.
* Teclistamab (TECVAYLI™) is a humanized IgG-4 PAA bispecific antibody designed to target the CD3 receptor complex on T cells and BCMA on B-lineage cells.
* Talquetamab (TALVEY™) is a humanized IgG-4 bispecific antibody designed to target the CD3 receptor complex on T cells and GPRC5D-expressing multiple myeloma (MM) cells This study will investigate the use of prophylactic tocilizumab or prophylactic dexamethasone to reduce the incidence and severity of CRS associated with teclistamab or talquetamab administration, to enable administration of the step-up dosing regimen of teclistamab or talquetamab in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age (or the higher legal age in the jurisdiction in which the study is taking place) at the time of informed consent
* Has documented diagnosis of MM according to the IMWG diagnostic criteria (Rajkumar 2011).
* Teclistamab or Talquetamab + Tocilizumab: has received 2 or more prior MM therapies including a PI, IMiD and CD38 antibody.
* Teclistamab + Oral Dexamethasone: has received 1 or more prior MM therapies including a PI, IMiD and/or CD38 antibody.
* Teclistamab or Talquetamab + Tocilizumab: has an ECOG performance status (Oken 1982) of 0 to 1.

Teclistamab + Oral Dexamethasone: has an ECOG performance status (Oken 1982) of 0 to 2.

* Measurable disease at screening, as assessed by local laboratory, defined by any of the following:

  * Serum M-protein level ≥0.5 g/dL; or
  * Urine M-protein level ≥200 mg/24 hours; or
  * Light chain MM without measurable M-protein in the serum or the urine: serum free light chain (sFLC) ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
  * For participants without measurable disease in the serum, urine, or involved FLC, presence of plasmacytomas (≥2 cm).
* Human immunodeficiency virus-positive participants are eligible if they meet all of the following:

  * No detectable viral load (i.e., <50 copies/mL) at screening
  * CD4+ count >300 cells/mm3 at screening
  * No acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within 6 months of screening
  * Receiving highly active antiretroviral therapy (HAART). Any changes in HAART due to resistance/progression should occur at least 3 months prior to enrollment. A change in HAART due to toxicity is allowed up to 4 weeks prior to enrollment.
* Adequate organ system function
* Body weight >35 kg.
* A participant of childbearing potential must have a negative highly sensitive serum (β-hCG) at screening and within 72 hours of the start of study treatment and must agree to further serum or urine pregnancy tests during the study.
* A participant must agree to abide by protocol defined contraceptive requirements for the duration of the study including avoiding donating gametes for specified period of time.
* A participant must sign an ICF indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.
* A participant is required to stay within 60 minutes of transportation to the site and remain in the company of a competent adult at all times until 48 hours following administration of all doses within the teclistamab step-up dosing schedules
* A participant is required to stay within 30 minutes of transportation to the site and remain in the company of a competent adult at all times until 48 hours following administration of all doses within the talquetamab step-up dosing schedule
* A participant must agree to carry the study participant identification wallet card at all times.
* A participant must comply with all the protocol requirement procedures, including measuring and recording of body temperature and blood oxygen saturation twice daily (≥8 hours apart) during the first 2 cycles of teclistamab or talquetamab treatment and coming to the study site for safety assessments.
* A participant and the accompanying competent adult must be made aware of the presenting sign sand symptoms of teclistamab- or talquetamab- associated toxicities, including but not limited to CRS, ICANS, infections, etc. The accompanying competent adult must watch the participant at all times for teclistamab- or talquetamab- associated toxicities, until 48 hours after the first treatment dose of teclistamab or talquetamab.

Exclusion Criteria:

* Has a rapidly progressing disease per investigator assessment.
* Has plasma cell leukemia (>2.0×10^9/L plasma cells by standard differential), Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary amyloid light-chain amyloidosis.
* Has known active CNS involvement or exhibits clinical signs of meningeal involvement of MM.
* Has risk factors for developing clinically significant TLS and requiring management with increased hydration, allopurinol, or rasburicase.
* Has myelodysplastic syndrome or active malignancies (ie, progressing or requiring treatment change in the last 12 months) other than RRMM. The only allowed exceptions are:

  * Any malignancy that was not progressing nor requiring treatment change in the last 12 months.
  * Malignancies treated within the last 12 months and considered at very low risk for recurrence:
  * Non-muscle invasive bladder cancer (solitary Ta-PUNLMP or low grade, <3 cm, no CIS).
  * Skin cancer (non-melanoma or melanoma).
  * Noninvasive cervical cancer.
  * Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, localized breast cancer and receiving antihormonal agents.
  * Localized prostate cancer (M0, N0) with a Gleason Score ≤7a, treated locally only (RP/RT/focal treatment).
  * Other malignancy that is considered at minimal risk of recurrence.
* Has Grade ≥3 hematologic AEs or Grade ≥3, clinically significant non-hematologic AEs.
* Has fever or active infection (bacterial, viral, or uncontrolled systemic fungal) at time of study enrollment.
* Has active autoimmune disease or a documented history of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing.
* Has clinically significant coagulopathy that would increase the risk of bleeding in the setting of cytopenia.
* Shows a deterioration in neurologic status, including mental status changes such as confusion or increased somnolence.
* Has psychiatric disorders (eg, alcohol or drug abuse), dementia, or altered mental status that would compromise the ability to provide informed consent or comply with the clinical protocol.
* History of stroke, transient ischemic attack or seizure within 6 months of signing ICF.
* Presence of the following cardiac conditions:

  * New York Heart Association stage III or IV congestive heart failure.
  * Myocardial infarction or CABG ≤6 months prior to enrollment.
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration.
  * History of severe non-ischemic cardiomyopathy.
  * Poorly controlled coronary artery disease and/or congestive heart failure.
  * Uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities.
* Has hepatitis B infection (ie, HBsAg or HBV-DNA positive). In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status.
* Has active hepatitis C infection as measured by positive HCV-RNA testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV-RNA positive) completed antiviral therapy and has undetectable HCV-RNA 12 weeks following the completion of therapy, the participant is eligible for the study.
* Has COPD with FEV1 <50% of predicted.
* Has eGFR <20 ml/min or is dependent on dialysis.
* Has other medical issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* For talquetamab arm only: Prior Grade 3 or higher CRS related to any T-cell redirection (e.g., CD-3 redirection technology or CAR-T cell therapy), or any prior GPRC5D-targeting therapy.
* Has received packed RBC or platelet transfusions within the last 7 days prior to dosing.
* Has contraindications to the use of tocilizumab or IVIG per local prescribing information.
* Has received live vaccine(s) within 1 month prior to screening or plans to receive live vaccines during the study.
* Has received live, attenuated vaccine(s) within 30 days before the first dose of teclistamab or talquetamab. Live, attenuated influenza vaccines are permitted as late as 30 days before the study treatment.
* Has received any non-cancer investigational intervention or used any non-cancer invasive investigational medical device within 14 days before the planned first dose of study treatment or received an investigational biological product within 14 days or 5 half-lives, whichever is shorter, before the planned study treatment, or is currently enrolled in an investigational study.
* History of anti-cancer therapy as follows, before the first dose of study drug:

  * Targeted therapy, epigenetic therapy, or treatment with an investigational drug or used an invasive investigational medical device within 21 days or at least 5 half-lives, whichever is less.
  * Monoclonal antibody treatment for MM within 21 days.
  * Cytotoxic therapy within 21 days.
  * PI therapy within 14 days.
  * Immunomodulatory agent therapy within 7 days.
  * Radiotherapy within 14 days or focal radiation within 7 days.
  * For teclistamab arms only: Prior Gene modified adoptive cell therapy (eg, chimeric antigen receptor modified [CAR]-T cells, NK cells, or BCMA therapy)
  * For talquetamab arm only: Prior CAR-T or BCMA bispecific antibody therapy are allowed with the appropriate wash-out period: 1) Gene modified adoptive cell therapy (eg, chimeric antigen receptor modified [CAR]-T cells, NK cells) within 3 months, or 2) BCMA therapies (antibody-drug conjugates and bispecific antibodies, etc) within 21 days or at least 5 half-lives, whichever is less.
* History of stem cell transplant:

  * An allogeneic stem cell transplant within 6 months. Participants who received an allogeneic transplant must be off all immunosuppressive medications for ≥42 days without signs of graft-versus-host disease.
  * An autologous stem cell transplant ≤12 weeks before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of CRS of any grade during the first two cycles | From first dose of teclistamab or talquetamab, from Day 1 first step-up dose to the end of Cycle 2 (each cycle is 28 days)
  Evaluate the overall incidence of CRS in the first 2 cycles after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.

SECONDARY OUTCOMES:
Incidence of recurrent CRS of any grade | From first dose of teclistamab or talquetamab, from Day 1 first step-up dose to the end of Cycle 2 (each cycle is 28 days)
  Evaluate the incidence of recurrent CRS either after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.
Incidence of CRS of any grade | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the incidence of CRS after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.
Incidence of recurrent CRS of any grade | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the incidence of recurrent CRS after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.
Incidence of Grade ≥2 CRS | From first dose of teclistamab or talquetamab, from Day 1 first step-up dose to the end of Cycle 2 (each cycle is 28 days)
  Evaluate the incidence of Grade ≥2 CRS based on American Society for Transplantation and Cellular Therapy (ASTCT) 2019 grading for CRS (Grade 1 to 5 with grade 5 defined as the worse outcome-Death) in the first 2 cycles after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.
Incidence of Recurrent Grade ≥2 CRS | From first dose of teclistamab or talquetamab, from Day 1 first step-up dose to the end of Cycle 2 (each cycle is 28 days)
  Evaluate the incidence of Grade ≥2 CRS based on American Society for Transplantation and Cellular Therapy (ASTCT) 2019 grading for CRS (Grade 1 to 5 with grade 5 defined as the worse outcome-Death) in the first 2 cycles after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.
Incidence of Grade ≥2 CRS | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the incidence of Grade ≥2 CRS based on American Society for Transplantation and Cellular Therapy (ASTCT) 2019 grading for CRS (Grade 1 to 5 with grade 5 defined as the worse outcome-Death) in the first 2 cycles and throughout the study after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.
Incidence of Recurrent Grade ≥2 CRS | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the incidence of Grade ≥2 CRS based on American Society for Transplantation and Cellular Therapy (ASTCT) 2019 grading for CRS (Grade 1 to 5 with grade 5 defined as the worse outcome-Death) in the first 2 cycles and throughout the study after a single dose of prophylactic tocilizumab given 2 to 4 hours prior to step-up dose 1 of teclistamab or talquetamab or after 3 doses of oral dexamethasone given after each step-up dose and the first full dose of teclistamab.
Incidence of Grade ≥3 and any grade infections | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the risk of Grade ≥3 and any grade infections throughout the study based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 (Grade 1 to 5 with grade 5 representing a worse outcome)
Incidence of All grade and Grade ≥3 neurotoxicity | From first dose of teclistamab or talquetamab, from Day 1 first step-up dose to the end of Cycle 2 (each cycle is 28 days)
  Evaluate neurotoxicity in the setting of prophylactic tocilizumab or prophylactic oral dexamethasone based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 (Grade 1 to 5 with grade 5 representing a worse outcome)
Incidence of All grade and Grade ≥3 ICANS | From first dose of teclistamab or talquetamab, from Day 1 first step-up dose to the end of Cycle 2 (each cycle is 28 days)
  Evaluate neurotoxicity including ICANS in the setting of prophylactic tocilizumab or prophylactic oral dexamethasone based on the American Society for Transplantation and Cellular Therapy (ASTCT) 2019 grading for ICANS (Grade 1 to 4 with grade 4 representing a worse outcome)
Incidence of All grade neutropenia and Grade ≥3 neutropenia | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate treatment-emergent neutropenia in the setting of teclistamab or talquetamab plus prophylactic tocilizumab or teclistamab plus prophylactic oral dexamethasone based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 (Grade 1 to 5 with grade 5 representing a worse outcome)
Incidence of all grade febrile neutropenia and Grade ≥3 febrile neutropenia | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate treatment-emergent febrile neutropenia in the setting of teclistamab or talquetamab plus prophylactic tocilizumab or teclistamab plus prophylactic oral dexamethasone based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 (Grade 1 to 5 with grade 5 representing a worse outcome)
Total length of each hospital stay | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the length of each hospital stay in the setting of teclistamab or talquetamab plus prophylactic tocilizumab or teclistamab plus prophylactic oral dexamethasone
Number of hospitalizations per participant | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the number of hospitalizations per participant, in the setting of teclistamab or talquetamab plus prophylactic tocilizumab or teclistamab plus prophylactic oral dexamethasone
Healthcare resource utilization in the outpatient setting | From first dose of teclistamab or talquetamab, from Day 1 first step-up dose to the end of Cycle 2 (each cycle is 28 days)
  Monitor the utilization of healthcare resources in the outpatient setting to mitigate the AEs associated with CRS/ICANS in the setting of teclistamab or talquetamab plus prophylactic tocilizumab or teclistamab plus prophylactic oral dexamethasone
Overall response rate (ORR) | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Overall response rate (ORR) will be defined as the proportion of participants who achieve a PR or better response according to the IMWG response criteria
Time to initial response (TTR) | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Time to initial response (TTR) will be defined as the time between the date of the first dose of teclistamab or talquetamab and the first efficacy evaluation that the participants have met all criteria for PR or better response according to the IMWG response criteria
Time to best response (TTBR) | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Time to best response (TTBR) will be defined as the time between the date of the first dose of teclistamab or talquetamab and the first efficacy evaluation that the participants have the best response according to the IMWG response criteria
Duration of response (DOR) | Day 1 of every 2 cycles from Cycle 1 Day 1 and up to approximately 12 months of teclistamab treatment or 6 months for talquetamab. (each cycle is 28 days)
  Duration of response (DOR) will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG response criteria
Time to next treatment (TTNT) | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Time to next treatment (TTNT) is defined as the time from the date of the first dose of teclistamab or talquetamab to the date of next treatment, or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Overall survival (OS) is defined as the time from the date of the first dose of teclistamab or talquetamab to the date of death, due to any cause.
Progression-free survival (PFS) | Day 1 of every 2 cycles From Cycle 1 Day 1 and up to approximately 12 months of teclistamab or 6 months for talquetamab treatment. (each cycle is 28 days)_
  Progression-free survival (PFS) is defined as the time from the date of the first dose of teclistamab or talquetamab, to the date of first documented disease progression, as defined in the IMWG response criteria, or death due to any cause, whichever occurs first.
Timing of each hospital stay | Up to 12 months of teclistamab or 6 months for talquetamab treatment
  Evaluate the timing of each hospital stay in the setting of teclistamab or talquetamab plus prophylactic tocilizumab or teclistamab plus prophylactic oral dexamethasone
Talquetamab Arm only: Number of participants who have had a change in health-related quality of life parameters, from baseline to end of treatment | Up to 6 months for talquetamab treatment
  Talquetamab Arm only: Assess health-related quality of life parameters related to overall health as well as specific impact of taste changes, xerostomia, dysphagia, oral mucositis, and other aspects of oral toxicity using EORTC-QLQ and Epstein taste scale
Talquetamab Arm only: Number of participants with oral toxicities | Up to 6 months for talquetamab treatment
  Talquetamab Arm only: Assess health-related quality of life parameters related to overall health as well as specific impact of taste changes, xerostomia, dysphagia, oral mucositis, and other aspects of oral toxicity using Epstein taste scale, PRO-CTCAE, STTA and SXI
Talquetamab Arm only: Number of patients with overall side effects | Up to 6 months for talquetamab treatment
  Talquetamab Arm only: Assess health-related quality of life parameters related to overall health as well as specific impact of taste changes, xerostomia, dysphagia, oral mucositis, and other aspects of oral toxicity using PGI-S and EORTC Q168/EORTC-IL46
Talquetamab Arm only: Rate of treatment-emergent dysgeusia, oral mucositis, dysphagia, and xerostomia | Up to 6 months for talquetamab treatment
  Talquetamab Arm only: To assess rate of treatment-emergent dysgeusia, oral mucositis, dysphagia, and xerostomia
Talquetamab Arm only: Time to first onset of treatment-emergent dysgeusia, oral mucositis, dysphagia, and xerostomia | Up 6 to months for talquetamab treatment
  Talquetamab Arm only: To assess time to first onset of treatment-emergent dysgeusia, oral mucositis, dysphagia, and xerostomia
Talquetamab Arm only: Duration of treatment-emergent dysgeusia, oral mucositis, dysphagia, and xerostomia | Up 6 to months for talquetamab treatment
  Talquetamab Arm only: To assess duration of treatment-emergent dysgeusia, oral mucositis, dysphagia, and xerostomia

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Forsberg, MD, Study Chair — SCRI Development Innovations, LLC
Locations (17):
- United States (17):
  - Arizona Oncology Associates, Tucson, Arizona
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Florida Cancer Specialists, Lake Mary, Florida
  - Maryland Oncology Hematology, Columbia, Maryland
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Virginia Oncology Associates, Elizabeth City, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - TriStar Bone Marrow Transplant, Nashville, Tennessee
  - Vanderbilt- Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology, Austin, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Blue Ridge Cancer Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No